CLINICAL TRIAL: NCT02919618
Title: Phase I/II Study of EP-guided Noninvasive Cardiac Radioablation for Treatment of Ventricular Tachycardia
Acronym: ENCORE-VT
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Principal Investigator, Phillip Cuculich, M.D., Washington University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201606081
Record Dates: First submitted 2016-09-28; First posted 2016-09-29 (Estimated); Results first posted 2019-09-10 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-07

CONDITIONS: Ventricular Tachycardia; Cardiomyopathy; Premature Ventricular Contractions
Keywords: Ventricular Tachycardia; Ablation; Noninvasive
MeSH Terms: conditions — Tachycardia, Ventricular; Cardiomyopathies; Ventricular Premature Complexes | interventions — Radiosurgery

STUDY DESIGN:
Intervention Model Description: Noninvasive Cardiac Radioablation, all subjects
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- stereotactic body radiotherapy (SBRT) (Experimental): Noninvasive SBRT will be delivered in a single fraction to a region of the heart determined by EP-guidance, using noninvasive electrical mapping combined with anatomic imaging.
  Interventions: Radiation: stereotactic body radiotherapy (SBRT)

INTERVENTIONS:
Radiation: stereotactic body radiotherapy (SBRT) — (Cardiac ablative radiotherapy)

SUMMARY:
Phase I/II Study of EP-guided Noninvasive Cardiac Radioablation (ENCORE) for Treatment of Ventricular Tachycardia

DETAILED DESCRIPTION:
Patients with Ventricular Tachycardia (VT) who have failed standard therapy (medicines, invasive catheter ablation) have limited options, with one-year survival below 20%. Preclinical data demonstrate that single fraction stereotactic body radiotherapy (SBRT) to discrete portions of the heart is feasible and may result in a reduction or elimination of VT. The efficacy may be further improved when guided by cardiac electrophysiologic (EP) testing. In total, the mapping and ablation proposed for this EP-guided Noninvasive Cardiac Radioablation (ENCORE) is a rapid and totally non-invasive method. Overall safety and early efficacy of ENCORE have not been rigorously studied in a prospective trial to-date. The purpose of this phase I/II study is to demonstrate the short-term safety and preliminary efficacy of ENCORE for patients with life-threatening, treatment-refractory VT.

ELIGIBILITY:
Inclusion Criteria:

1. DOCUMENTED VT:

   1. Patient must have documented sustained monomorphic ventricular tachycardia as documented on either a 12-lead ECG or intracardiac ICD interrogation

      - OR-
   2. Monomorphic PVCs documented on a 12-lead ECG.
2. ANTIARRHYTHMIC MEDICATION: Patient must have failed or become intolerant to at least one antiarrhythmic medication (amiodarone, sotalol, or mexiletine).

   -AND-
3. CATHETER ABLATION: Patient must have failed at least one invasive catheter ablation procedure, or have a contraindication to a catheter ablation procedure (e.g., LV thrombus, severe pulmonary disease), or have VT thought to arise from a protected location (e.g., epicardial VT with history of previous cardiac surgery).
4. MINIMUM VT BURDEN: Patient must have either:

   1. At least 3 VT episodes (sustained VT, ICD ATP or ICD shock) over previous 6 months prior to enrollment -OR-
   2. >20% PVC burden with a cardiomyopathy (LVEF<50%)
5. Patient must be deemed medically fit for stereotactic body radiation therapy by the treating physician.
6. Patient must be > 18 years old.
7. Patient must be able to understand and be willing to sign an IRB approved written informed consent document.

   -

Exclusion Criteria:

1. Patient must not have past history of radiotherapy within the projected treatment field.
2. Advanced symptomatic heart failure as defined as NYHA Class IV heart failure (inotrope dependent and/or current left-ventricular assist device (LVAD))
3. Polymorphic VT or ventricular fibrillation (VF) as a clinical heart rhythm (as determined by 12-lead ECG and/or ICD interrogation).
4. More than 3 distinct clinical VT morphologies observed (ECG or ICD interrogation or invasive EP study) OR more than 5 distinct induced VT morphologies during ECGI testing.
5. Advanced myocardial scar substrate that would require stereotactic delivery to a target volume deemed unsafe by the treating physician.
6. Unlikely to live 12 months, in the absence of VT, as best based on clinical judgment by the treating and enrolling physicians.
7. Patient must not be pregnant and/or breastfeeding and must have a negative pregnancy test within 14 days of study entry.

   -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2018-07-23 (Actual); Study Completion 2024-01-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Phillip Cuculich, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Yes
Open sharing at the time of publication of results
Supporting Information: Study Protocol

REFERENCES:
- [Derived] Robinson CG, Samson PP, Moore KMS, Hugo GD, Knutson N, Mutic S, Goddu SM, Lang A, Cooper DH, Faddis M, Noheria A, Smith TW, Woodard PK, Gropler RJ, Hallahan DE, Rudy Y, Cuculich PS. Phase I/II Trial of Electrophysiology-Guided Noninvasive Cardiac Radioablation for Ventricular Tachycardia. Circulation. 2019 Jan 15;139(3):313-321. doi: 10.1161/CIRCULATIONAHA.118.038261. PMID 30586734

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Twenty-one patients were consented between July 11, 2016 and December 20, 2017. These patients were evaluated as either inpatient or outpatient. Once patients met initial enrollment criteria, screening procedures were conducted to determine if the patient was eligible for SBRT.
Pre-assignment Details: Nineteen patients were consented, screened, and deemed eligible for SBRT.
  Two additional patients signed consent and went through screening procedures; however, were later deemed ineligible to obtain SBRT.
Groups:
- Patients Overall Who Received SBRT: Noninvasive Stereotactic Body Radiotherapy (SBRT) will be delivered in a single fraction to a region of the heart determined by EP-guidance, using noninvasive electrical mapping combined with anatomic imaging.
  Stereotactic Body Radiotherapy (SBRT): (Cardiac ablative radiotherapy)
Period: Overall Study
Arm/Group | Patients Overall Who Received SBRT
Started | 19
Primary Safety Endpoint (</=90 Days) (Phase 1 - Defined by a </=20% rate of SAEs using CTCAE v4.0 criteria.) | 19
Primary Efficacy Endpoint (6 Months) (Phase 2 - Number of subjects with a reduction in ICD therapies 6mo before and 6mo post-SBRT.) | 18
Completed | 18
Not Completed | 1
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Groups:
- Patients Overall Who Received SBRT: Noninvasive SBRT will be delivered in a single fraction to a region of the heart determined by EP-guidance, using noninvasive electrical mapping combined with anatomic imaging.
  Stereotactic Body Radiotherapy (SBRT): (Cardiac ablative radiotherapy)
Arm/Group | Patients Overall Who Received SBRT
Number analyzed (Participants) | 19
Age, Continuous [Median (Full Range); unit: years] | 66 [49 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 17
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 17
  More than one race | 0
  Unknown or Not Reported | 0
BMI [Median (Full Range); unit: kg/m^2] | 33.0 [24.3 to 48.6]
Age-Adjusted Charlson Comorbidity Index [Median (Full Range); unit: Score] — The Charlson Comorbidity Index predicts 10-year survival in patients with multiple comorbidities. The Charlson Comorbidity Index scale ranges from 0 (no comorbidities) to 37 (all comorbidities in equation). The score is then adjusted based on the age of the patient, adding 0 to 4 points to the Charlson Comorbidity Index score, thus providing the Age-Adjusted Charlson Comorbidity Index.
  Score | 4 [2 to 13]
Type of Cardiomyopathy [Count of Participants; unit: Participants]
  Ischemic Cardiomyopathy | 11
  Nonischemic Cardiomyopathy | 8
Type of Nonischemic Cardiomyopathy [Count of Participants; unit: Participants] — Population: Based on the number of patients enrolled with nonischemic cardiomyopathy (8/19).
  Participants
    number analyzed (Participants) | 8
    Idiopathic | 5
    Myocarditis (Chronic) | 2
    Valvular | 1
New York Heart Association (NYHA) Class [Count of Participants; unit: Participants] — NYHA Class I: No limitation of physical activity. Ordinary physical activity does not cause undue fatigue, palpitation, dyspnea; NYHA Class II: Slight limitation of physical activity. Comfortable at rest. Ordinary physical activity results in fatigue, palpitation, dyspnea; NYHA Class III: Marked limitation of physical activity. Comfortable at rest. Less than ordinary activity causes fatigue, palpitation, dyspnea; NYHA Class IV: Unable to carry on any physical activity without discomfort. Symptoms of heart failure at rest. If any physical activity is undertaken, discomfort increases.
  Participants
    NYHA I | 1
    NYHA II | 4
    NYHA III | 10
    NYHA IV | 4
Left Ventricular Ejection Fraction [Median (Full Range); unit: Percentage of Ejection Fraction] | 25 [15 to 58]
Number of Previous Catheter Ablations [Median (Full Range); unit: Invasive Procedures] | 1 [0 to 4]
Total Number of Prior Catheter Ablation Approaches [Number; unit: Invasive Ablation Approaches]
  Endocardial | 25
  Epicardial | 4
Study Eligibility Criteria [Count of Participants; unit: Participants]
  Incessant Ventricular Tachycardia (VT) | 2
  VT Storm (>3 episodes of VT in 24 hours) | 10
  ICD Therapies (>3 shocks or ATP in 6 months) | 5
  PVC-Related Cardiomyopathy | 2
Device [Count of Participants; unit: Participants]
  Single- or Dual-Chamber ICD | 8
  Biventricular ICD | 10
  No Device | 1
Current Antiarrhythmic Drugs [Number; unit: Count of Participants]
  >1 Antiarrhythmic Drug at Baseline | 11
  High-Dose Amiodarone (>/=300mg per day) | 10
  Low-Dose Amiodarone (<300mg per day) | 2
  Class III (excluding amiodarone) | 7
  Class I | 11
Other Medications [Number; unit: Count of Participants]
  Beta Blocker | 18
  Angiotensin Converting Enzyme Inhibitor | 10
  Angiotensin Receptor Blocker | 7
  Oral Anticoagulation | 14
Variable [Number; unit: Count of Participants]
  Chronic Obstructive Pulmonary Disease/Emphysema | 4
  Diabetes Mellitus, Type II | 7
  Hypertension | 10
  Chronic Kidney Disease (Stage >/=3) | 9

OUTCOME MEASURES:

1. Primary Outcome: Number of Serious Adverse Events
Description: Demonstrate acute (≤ 90 days) safety of noninvasive stereotactic cardiac ablation radiotherapy (ENCORE). The primary safety endpoint is defined by a ≤ 20% rate of serious adverse events (SAEs) using CTCAE v4.0 criteria that are possibly/probably/definitely related to study treatment, based on previously published data for expected invasive catheter-based VT-ablation procedures.
Time Frame: < or = 90 days
Population: Analysis is based on number of SAE events that occurred in 19 participants within 90 days after SBRT.
Measure: Number; unit: Events
Groups:
- Number of Events: Number of serious adverse events that occurred.
Arm/Group | Number of Events
Number analyzed (Participants) | 19
Events
  Grade 3 treatment-related SAE | 2
  Grade 4 treatment-related SAE | 0
  Grade 5 treatment-related SAE | 0
  Grade 5 SAE (not treatment-related) | 1

2. Primary Outcome: Number of Participants With Reduction in Ventricular Tachycardia (VT) Burden
Description: Primary efficacy endpoint is defined by the number of subjects with a reduction in VT burden comparing the period six months before ENCORE treatment to the six months after ENCORE treatment as adjudicated by continuous ICD monitoring (number of ATP and ICD shocks and sustained (>30 second) nontreated slow VT). There will be a six-week "blanking period" after therapy to allow for ablation effect. For patients with PVC-induced cardiomyopathy, the primary efficacy will be any reduction in PVC burden based on ambulatory heart monitors.
Time Frame: 12 months (6mo prior to and 6mo post SBRT)
Population: Percent reduction of VT episodes or PVC burden 6 months post-SBRT compared to 6 months prior to SBRT.
  Patients who were alive at 6 months were evaluated comparing ICD treatments or PVC burden 6 months before and 6 months post-SBRT.
Measure: Count of Participants; unit: Participants
Groups:
- Patients With ICD-treated VT Indication: Sixteen evaluable patients out of the overall 18 patients alive at 6 months who were enrolled with an ICD-treated VT indication.
- Patients With PVC-Related Cardiomyopathy Indication: Two evaluable patients out of the overall 18 patients alive at 6 months who were enrolled with a PVC indication.
Arm/Group | Patients With ICD-treated VT Indication | Patients With PVC-Related Cardiomyopathy Indication
Number analyzed (Participants) | 16 | 2
Participants | 15 | 2

3. Secondary Outcome: Overall Survival
Description: Determine six-month and twelve-month survival (overall mortality endpoint) after treatment with ENCORE.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Groups:
- 6 Month Overall Survival: Overall survival at the 6 month post-SBRT time point of all 19 patients enrolled.
- 12 Month Overall Survival: Overall survival at the 12 month post-SBRT time point of the 18 remaining patients from the 6 month time point.
Arm/Group | 6 Month Overall Survival | 12 Month Overall Survival
Number analyzed (Participants) | 19 | 18
Participants | 18 | 13

4. Secondary Outcome: Number of Adverse Events That Are Possibly/Probably/Definitely Related to Study Treatment
Description: Toxicities that occur after treatment, but are not acutely ascribed to treatment that are possibly/probably/definitely related to study treatment, based on previously published data for expected invasive catheter-based VT-ablation procedures, using the CTCAE v4.0 criteria.
Time Frame: 90 days to 12 months
Population: Analysis is based on number of AE events that occurred in 18 participants >90 days to 365 days post-SBRT.
Measure: Number; unit: Number of Events
Groups:
- Number of Events: Number of adverse events that occurred.
Arm/Group | Number of Events
Number analyzed (Participants) | 19
Number of Events
  Grade 1 Possibly Related AE | 15
  Grade 1 Probably Related AE | 1
  Grade 2 Possibly Related AE | 9
  Grade 2 Probably Related AE | 1
  Grade 2 Definitely Related AE | 1
  Grade 3 Possibly Related AE | 20
  Grade 4 Possibly Related AE | 1
  Grade 5 Possibly Related AE | 1

5. Secondary Outcome: Health Related Quality of Life (HRQOL)
Description: The 36-Item Short Form Survey (SF-36) is a set of generic, coherent, and easily administered quality of life measures that rely on patient self-reporting. The SF-36 evaluates 8 domains: physical functioning, bodily pain, role limitations due to physical health problems, role limitations due to personal or emotional problems, emotional well-being, social functioning, energy/fatigue, and general health perceptions. Scale values for each domain range from 0 to 100 where the higher score defines a more favorable health state.
Time Frame: 6 week, 6 month, 12 month
Measure: Mean (Full Range); unit: Scores on a Scale
Groups:
- Baseline: Baseline mean scores for all 18 evaluable patients at the 6 week time point.
- 6 Week: 6 week mean scores for all 18 evaluable patients at the 6 week time point.
- 6 Month: 6 month mean scores for all 16 evaluable patients at the 6 month time point. 2 patients did not return the SF-36 survey for the 6 month follow up.
- 12 Month: 12 month mean scores for all 13 evaluable patients at the 12 month time point. 5 patients had expired prior to the 12 month time point.
Arm/Group | Baseline | 6 Week | 6 Month | 12 Month
Number analyzed (Participants) | 18 | 18 | 16 | 13
Scores on a Scale
  Social Functioning | 64 [25 to 100] | 70 [13 to 100] | 87 [50 to 100] | 72 [38 to 100]
  General Health | 44 [10 to 85] | 52 [15 to 95] | 49 [6 to 90] | 54 [15 to 85]
  Health Change | 28 [0 to 75] | 61 [25 to 100] | 77 [0 to 100] | 65 [0 to 100]

6. Secondary Outcome: Number of Participants With a 50% Reduction in Ventricular Tachycardia (VT) Burden
Description: Evaluate stricter efficacy endpoint of ENCORE treatment, as defined by number of patients who have had 50% reduction in any VT therapies (ATP or ICD shocks or sustained (>30sec) nontreated slow VT) after ENCORE treatment (6 months before vs. 6 months after treatment, with a 6 week blanking period immediately after treatment). For patients with PVC-induced cardiomyopathy, the stricter efficacy will be >50% reduction in PVC burden based on ambulatory heart monitors.
Time Frame: 6 months
Population: One patient was excluded because they expired prior to the outcome measure time frame.
Measure: Count of Participants; unit: Participants
Arm/Group | Patients Overall Who Received SBRT
Number analyzed (Participants) | 18
Participants | 17

7. Secondary Outcome: Number of Participants With a 95% Reduction in Ventricular Tachycardia (VT) Burden
Description: Evaluate strictest efficacy endpoint of ENCORE treatment, as defined by number of patients who have had 95% reduction in any VT (ATP or ICD shocks or sustained (>30 sec) slow VT) after ENCORE treatment (6 months before vs. 6 months after treatment, with a 6 week blanking period immediately after treatment). For patients with PVC-induced cardiomyopathy, the strictest efficacy will be abolition of PVC burden (<1%) based on ambulatory heart monitors.
Time Frame: 6 months
Population: One patient was excluded because they expired prior to the outcome measure time frame.
Measure: Count of Participants; unit: Participants
Arm/Group | Patients Overall Who Received SBRT
Number analyzed (Participants) | 18
Participants | 11

8. Secondary Outcome: Number of Participants With Reduction in ICD Shocks and LVEF Improvement
Description: Evaluate the most clinically useful efficacy endpoint of ENCORE treatment, namely, number of patients with reduction specifically in ICD shocks (6 months before vs. 6 months after treatment, with a 6 week blanking period immediately after treatment). For patients with PVC-induced cardiomyopathy, the most clinically useful efficacy will be improvement in cardiac function in the setting of any improvement in PVC burden.
Time Frame: 6 months
Population: One patient was excluded because they expired prior to the outcome measure time frame.
Measure: Count of Participants; unit: Participants
Arm/Group | Patients Overall Who Received SBRT
Number analyzed (Participants) | 18
Participants | 13

9. Secondary Outcome: Number of Participants With Reduction in Ventricular Tachycardia (VT) Therapies Between 6 and 12 Months
Description: Evaluate longer-term durability endpoint of ENCORE treatment, as defined by number of patients with reduction in VT therapies (ATP or ICD shock or sustained (>30 sec) slow VT and ICD shock alone) during the early phase (treatment to 6 months, with 6 week blanking period) vs. the late phase (6 months to 1 year). For patients with PVC-induced cardiomyopathy, the longer-term durability efficacy will be persistence of any reduction in PVC burden based on ambulatory heart monitors during early phase vs. late phase.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Patients Overall Who Received SBRT
Number analyzed (Participants) | 18
Participants | 16

ADVERSE EVENTS:
Time Frame: Adverse Event data provided was obtained for all participants up to 1 year post-SBRT for last treated participant.
Arm/Group | Patients Overall Who Received SBRT
All-Cause Mortality (participants affected / at risk) | 8/19
Serious Adverse Events (participants affected / at risk) | 15/19
Other Adverse Events (participants affected / at risk) | 19/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Patients Overall Who Received SBRT (N=19)
Acidosis (Metabolism and nutrition disorders) | 1
Acute Kidney Injury (Renal and urinary disorders) | 2
Anemia (Blood and lymphatic system disorders) | 1
Atrial Fibrillation (Cardiac disorders) | 1
Cardiac Arrest (Cardiac disorders) | 3
Cholecystitis (Hepatobiliary disorders) | 1
Cognitive Disturbance (Nervous system disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Diarrhea (Gastrointestinal disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2
Flushing (Vascular disorders) | 1
Gastric Hemorrhage (Gastrointestinal disorders) | 1
Heart Failure (Cardiac disorders) | 6
Hematoma (Vascular disorders) | 1
Hepatic Failure (Hepatobiliary disorders) | 1
Hypertension (Vascular disorders) | 1
Hypotension (Vascular disorders) | 3
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2
Intraoperative Cardiac Injury (Injury, poisoning and procedural complications) | 1
Multi-organ Failure (General disorders) | 1
Other - Accident (General disorders) | 1
Other - Chemical Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 — Amiodarone Induced
Other - Chest Pain NOS (Cardiac disorders) | 2
Other - Pneumonia (Respiratory, thoracic and mediastinal disorders) | 2
Other - ICD Lead Fracture (Cardiac disorders) | 1
Palpitations (Cardiac disorders) | 1
Pericardial Effusion (Cardiac disorders) | 2
Pericarditis (Cardiac disorders) | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 2
Retroperitoneal Hemorrhage (Gastrointestinal disorders) | 1
Urinary Tract Infection (Infections and infestations) | 1
Ventricular Fibrillation (Cardiac disorders) | 1
Ventricular Tachycardia (Cardiac disorders) | 9
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Patients Overall Who Received SBRT (N=19)
Abdominal Pain (Gastrointestinal disorders) | 2
Acute Coronary Syndrome (Cardiac disorders) | 1
Acute Kidney Injury (Renal and urinary disorders) | 1
Agitation (Psychiatric disorders) | 1
Alanine Aminotransferase Increased (Investigations) | 1
Alkaline Phosphatase Increased (Investigations) | 1
Allergic Reaction (Immune system disorders) | 1 — Due to MRI contrast
Ankle Fracture (Injury, poisoning and procedural complications) | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 1
Aspartate Aminotransferase Increased (Investigations) | 1
Atrial Fibrillation (Cardiac disorders) | 2
Back Pain (Musculoskeletal and connective tissue disorders) | 4
Blood Bilirubin Increased (Investigations) | 1
Chest Wall Pain (Musculoskeletal and connective tissue disorders) | 1
Chills (General disorders) | 1
Cholecystitis (Hepatobiliary disorders) | 1
Colitis (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 3
Cyst (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Dizziness (Nervous system disorders) | 9
Dysesthesia (Nervous system disorders) | 3
Dyspepsia (Gastrointestinal disorders) | 6
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 8
Ear Pain (Ear and labyrinth disorders) | 1
Fatigue (General disorders) | 12
Fracture (Injury, poisoning and procedural complications) | 1
Headache (Nervous system disorders) | 2
Heart Failure (Cardiac disorders) | 8
Hematoma (Vascular disorders) | 1
Hematuria (Renal and urinary disorders) | 2
Hyperglycemia (Metabolism and nutrition disorders) | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2
Hypersomnia (Nervous system disorders) | 1
Hypertension (Vascular disorders) | 1
Hypotension (Vascular disorders) | 8
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Malaise (General disorders) | 1
Mitral Valve Disease (Cardiac disorders) | 1 — Progression of existing mitral regurgitation
Nausea (Gastrointestinal disorders) | 6
Other - Chest Pain NOS (Cardiac disorders) | 8
Other - Congestive Gastropathy (Gastrointestinal disorders) | 1
Other - Dark Stools (Gastrointestinal disorders) | 1
Other - Dysuria (Renal and urinary disorders) | 1
Other - Gastroenteritis (Gastrointestinal disorders) | 1
Other - Influenza (Respiratory, thoracic and mediastinal disorders) | 1
Other - Nephrolithiasis (Renal and urinary disorders) | 1
Other - Pneumonia (Respiratory, thoracic and mediastinal disorders) | 2
Other - Polydipsia (Gastrointestinal disorders) | 1
Other - Radiation Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2
Other - Shoulder Pain (Musculoskeletal and connective tissue disorders) | 1
Other - Tendon Rupture (Musculoskeletal and connective tissue disorders) | 1
Palpitations (Cardiac disorders) | 1
Paresthesia (Nervous system disorders) | 1
Pericardial Effusion (Cardiac disorders) | 5
Pericarditis (Cardiac disorders) | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 2
Pleuritic Pain (Respiratory, thoracic and mediastinal disorders) | 1
Presyncope (Nervous system disorders) | 1
Pulmonary Edema (Respiratory, thoracic and mediastinal disorders) | 1
Retroperitoneal Hemorrhage (Gastrointestinal disorders) | 1
Seizure (Nervous system disorders) | 1
Sepsis (Infections and infestations) | 1
Sinus Tachycardia (Cardiac disorders) | 1
Sinusitis (Infections and infestations) | 1
Spacticity (Nervous system disorders) | 1
Stomach Pain (Gastrointestinal disorders) | 1
Syncope (Nervous system disorders) | 1
Testicular Pain (Reproductive system and breast disorders) | 1
Thromboembolic Event (Vascular disorders) | 1
Tremors (Nervous system disorders) | 1 — Amiodarone Induced
Upper Respiratory Infection (Infections and infestations) | 3
Urinary Tract Infection (Infections and infestations) | 1
Ventricular Fibrillation (Cardiac disorders) | 1
Vomiting (Gastrointestinal disorders) | 5
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-09-26): https://cdn.clinicaltrials.gov/large-docs/18/NCT02919618/Prot_SAP_000.pdf